CLINICAL TRIAL: NCT06932081
Title: Adult Congenital Heart Disease International EValuation of the Effectiveness of SGLT2i (ACHIEVE-SGLT2i) Registry
Brief Title: Adult Congenital Heart Disease International EValuation of the Effectiveness of SGLT2i Registry
Acronym: ACHIEVE-SGLT2i
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, aegorova, Principal Investigator, Leiden University Medical Center
Other Study IDs: 2022-068
Record Dates: First submitted 2025-03-02; First posted 2025-04-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Adult Congenital Heart Disease; Congenital Heart Disease; Systemic Right Ventricle; Transposition of the Great Arteries; Congenitally Corrected Transposition of the Great Arteries; Fontan; Single Ventricle; Tetralogy of Fallot (TOF)
Keywords: adult congenital heart disease; ACHD; congenital heart disease; CHD; sodium-glucose cotransporter 2 inhibitors; SGLT2i; SGLT2; heart failure; HF; transposition of the great arteries; TGA; systemic right ventricle; sRV; Fontan; single ventricle; tetralogy of fallot; ToF
MeSH Terms: conditions — Heart Defects, Congenital; Transposition of Great Vessels; Congenitally Corrected Transposition of the Great Arteries; Univentricular Heart; Tetralogy of Fallot; Heart Failure | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ACHD patients treated with SGLT2i: All participants included in the registry have to have a congenital heart defect, be ≥ 18 years old, and receive (or have received) treatment with SGLT2i.
  Interventions: Drug: SGLT2 inhibitors

INTERVENTIONS:
Drug: SGLT2 inhibitors — Treatment with any type and dose of sodium-glucose cotransporter 2 inhibitor.

SUMMARY:
This real-world, international registry aims to evaluate the current experience with sodium-glucose cotransporter 2 inhibitors (SGLT2i) in adult congenital heart disease (ACHD) patients by investigating the prescription patterns, safety, tolerability, and potential beneficial effects on heart failure-related outcomes.

DETAILED DESCRIPTION:
In the adult congenital heart disease (ACHD) population, heart failure currently represents the main cause of morbidity and mortality. The etiology of ACHD-related heart failure is heterogenous, and there is limited evidence for pharmacological treatment options for this population.

Sodium-glucose cotransporter 2 inhibitors (SGLT2i) are a novel pillar in the treatment of conventional LV heart failure. SGLT2i have been shown to reduce the risk of worsening heart failure and cardiovascular-related death in patients with LV heart failure.

While the exact mechanisms of action are still to be elucidated, SGLT2i seem to address heart failure by targeting several pathways. These include but are not limited to; a decrease in renin-angiotensin and sympathetic nervous system activation, a decrease in pressure overload-induced myocardial fibrosis, reverse cardiac remodeling, and improvement in myocardial energetics.

Given the compelling evidence on the effectiveness of SGLT2i over a broad range of cardiac dysfunction and initial promising reports of its utilization in the field of ACHD, SGLT2i deserve further exploration in the group of ACHD patients.

This real-world, international registry aims to evaluate the current experience with SGLT2i in ACHD patients by investigating the prescription patterns, safety, tolerability, and potential beneficial effects on heart failure-related outcomes.

Project design:

Data of all ACHD patients who were started on an SGLT2i will be collected in a real-world, international registry. Only data resulting from routine clinical care will be collected from the electronic health records at the participating centers, and participants will not undergo any interventions for this project. Data will be collected from 1 year before starting with the SGLT2i to most recent follow-up after starting with the SGLT2i, to evaluate if SGLT2i therapy halts the progression of clinical deterioration in ACHD patients with heart failure and can improve heart failure-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart defect.
* Age ≥ 18 years.
* Initiated on treatment with an SGLT2i.

Exclusion Criteria:

- No consent for data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years) with congenital heart disease who have been treated with an SGLT2i are eligible for inclusion in the registry.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Prescription patterns | Baseline information.
  The primary outcome of this registry is an overview of the prescription patterns of SGLT2i in the ACHD population.

SECONDARY OUTCOMES:
Side effects [Safety and Tolerability] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Incidence and specification of any experienced side effects.
SGLT2i-related complications [Safety and Tolerability] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Incidence and specification of any SGLT2i-related complications.
SGLT2i discontinuation [Safety and Tolerability] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Incidence of any discontinuation of SGLT2i (including reason for discontinuation).
Mortality [Safety and Tolerability] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Mortality and documentation of cause of death.
Admissions [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Documentation of number of hospitalizations, including number of heart failure-related hospitalizations and number of urgent heart failure visits.
Clinical parameters - weight [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on weight (kg)
Clinical parameters - systolic blood pressure [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on systolic blood pressure (mmHg)
Clinical parameters - diastolic blood pressure [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on diastolic blood pressure (mmHg)
Clinical parameters - heart rate [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on heart rate (beats per minute)
Clinical parameters - saturation [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on oxygen saturation (%)
Laboratory parameters - sodium [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on serum sodium (mmol/L)
Laboratory parameters - potassium [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on serum potassium (mmol/L)
Laboratory parameters - creatinine [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on serum creatinine (µmol/L)
Laboratory parameters - eGFR [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on estimated glomerular filtration rate (eGFR, ml/min/1.73m2)
Laboratory parameters - NT-proBNP [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on serum NT-proBNP (ng/L)
Laboratory parameters - glucose [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on serum glucose (mmol/L)
Laboratory parameters - HbA1c [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on serum HbA1c (mmol/mol Hb)
Transthoracic echocardiography - LV function [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on systolic left ventricular (LV) function (categorical: good, mildly reduced, moderately reduced, severely reduced function)
Transthoracic echocardiography - LV GLS [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on LV global longitudinal strain (GLS, %) assessed with transthoracic echocardiography
Transthoracic echocardiography - LV FAC [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on LV fractional area change (FAC, %) assessed with transthoracic echocardiography
Transthoracic echocardiography - RV function [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on systolic right ventricular (RV) function (categorical: good, mildly reduced, moderately reduced, severely reduced function) assessed with transthoracic echocardiography
Transthoracic echocardiography - RV GLS [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on RV GLS (%) assessed with transthoracic echocardiography
Transthoracic echocardiography - RV FAC [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on RV FAC (%) assessed with transthoracic echocardiography
Transthoracic echocardiography - RV S' [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on RV S' (cm/s) assessed with transthoracic echocardiography
Transthoracic echocardiography - TAPSE [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on tricuspid annular plane systolic excursion (TAPSE, mm) assessed with transthoracic echocardiography
Exercise parameters - 6MWT [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on exercise parameter 6-minute walk test (6MWT, meters)
Exercise parameters - maximum performance [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on maximum performance (Watt) with bicycle ergometry.
Exercise parameters - validity [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on validity (%-predicted of the maximum performance) with bicycle ergometry.
Exercise parameters - VO2 max [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on VO2 max (mL/kg/min) with bicycle ergometry.
Exercise parameters - %-predicted VO2 max [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the longitudinal effect of SGLT2i on %-predicted of VO2 max (% of the VO2 max) with bicycle ergometry.
Concomitant medication changes [Heart Failure-related Efficacy] | From enrollment through study completion, with an average follow-up duration of 1 year.
  Evaluation of the concomitant changes in other heart failure pharmacotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia D. Egorova, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (10):
- United States (3):
  - Johns Hopkins University, Baltimore, Maryland
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Mount Sinai Fuster Heart Hospital, New York, New York
- Netherlands (3):
  - Leiden University Medical Center (LUMC), Leiden, South Holland
  - Amsterdam University Medical Center, Amsterdam
  - University Medical Center Utrecht, Utrecht
- Zan Mitrev Clinic, Skopje, North Macedonia
- United Kingdom (3):
  - University Hospital of Wales, Cardiff
  - Golden Jubilee University National Hospital, Glasgow
  - Barts Heart Centre, London

REFERENCES:
- [Background] Neijenhuis RML, MacDonald ST, Zemrak F, Mertens BJA, Dinsdale A, Hunter A, Walker NL, Swan L, Reddy S, Rotmans JI, Jukema JW, Jongbloed MRM, Veldtman GR, Egorova AD. Effect of Sodium-Glucose Cotransporter 2 Inhibitors in Adults With Congenital Heart Disease. J Am Coll Cardiol. 2024 Apr 16;83(15):1403-1414. doi: 10.1016/j.jacc.2024.02.017. Epub 2024 Mar 25. PMID 38530688
- [Background] Neijenhuis RML, Nederend M, Jongbloed MRM, Kies P, Rotmans JI, Vliegen HW, Jukema JW, Egorova AD. The potential of sodium-glucose cotransporter 2 inhibitors for the treatment of systemic right ventricular failure in adults with congenital heart disease. Front Cardiovasc Med. 2023 Jun 26;10:1093201. doi: 10.3389/fcvm.2023.1093201. eCollection 2023. PMID 37435053
- [Background] Egorova AD, Nederend M, Tops LF, Vliegen HW, Jongbloed MRM, Kies P. The first experience with sodium-glucose cotransporter 2 inhibitor for the treatment of systemic right ventricular failure. ESC Heart Fail. 2022 Jun;9(3):2007-2012. doi: 10.1002/ehf2.13871. Epub 2022 Mar 30. PMID 35355435